CLINICAL TRIAL: NCT03899350
Title: The Influencing Factors and Prediction Model of Poor Prognosis of Spontaneous Intraparenchymal Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDSJWKICH
Record Dates: First submitted 2019-01-07; First posted 2019-04-02 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Spontaneous Intracranial Hemorrhage; Spontaneous Intraparenchymal Cerebral Hemorrhage; Spontaneous Cerebellar Haemorrhage
Keywords: Treatment Efficacy; Intraparenchymal Hemorrhage; Surgery; Outcome; Prediction Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spontaneous Supratentorial Intracerebral Haemorrhage: Participants with spontaneous supratentorial intracerebral haemorrhage.
  Interventions: Other: No intervention
- Spontaneous Intracerebellar Hemorrhage: Participants with spontaneous intracerebellar hemorrhage.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study was designed to explore the influencing factors of spontaneous intraparenchymal hemorrhage's prognosis and develop predictive models for poor prognosis by establishing a cohort of spontaneous intraparenchymal hemorrhage (including both of the supratentorial intracerebral hemorrhage and cerebellar hemorrhage), and analyzing the correlation between collected variables and patients' outcomes.

DETAILED DESCRIPTION:
Spontaneous intracranial hemorrhage is an important type of cerebrovascular disease. The disease has an acute onset, a serious condition, and a high mortality rate. Besides, the survivors always live with severe neurological dysfunction. It is essential to determine the influencing factors of poor prognosis, estimate patient's condition and predict the prognosis timely.

This study consists of two parts. The first part establishes a cohort of spontaneous intraparenchymal hemorrhage (including both of the supratentorial intracerebral hemorrhage and cerebellar hemorrhage), and analyzes the influence of different factors, such as surgical methods, on the prognosis. In the second part, a nested case-control study nested in this cohort will be established to analyse the influence of some other factors. The biological specimens are tested. The collected data were analysed to find out the risk factors of poor prognosis and establish a predictive model.

Recruitment and follow-up of the participants is expected to continue after the initial goal is achieved. As a large sample database of intracranial hemorrhage, this cohort will provide more research data for the future exploration of more clinical problems.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80；
2. Diagnosed with spontaneous intraparenchymal hemorrhage (both of the supratentorial intracerebral hemorrhage and cerebellar hemorrhage) by Computed Tomography;
3. Admitted within 24h of ictus；
4. Did not undertake treatment before enrollment;
5. Informed consent to participate in the study.

Exclusion Criteria:

1. The hemorrhage caused by tumor, arteriovenous malformation, aneurysm or coagulopathy；
2. Concurrent traumatic brain injury；
3. Multiple intracerebral hemorrhage；
4. Undertake any surgery after onset in other hospital；
5. Refuse the treatment after admission;
6. History of craniocerebral surgery；
7. Known advanced demential or disability before onset；
8. Any concurrent serious illness that would interfere with the safety assessments including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, and hematologic disease;
9. Confirmed malignant disease or life expectancy less than 6 months due to comorbid diseases;
10. Concurrent serious infectious disease (HIV, tuberculosis etc.)
11. Concurrent coagulation disorders or having taken anti-platelet or anticoagulant drugs;
12. With indications of terminal brain hernia
13. Pregnant or lactating females；
14. Participation in another simultaneous trial of intracerebral hemorrhage treatment；
15. Patients/relatives refuse to be followed up。

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All of the spontaneous intraparenchymal hemorrhage (both of the supratentorial intracerebral hemorrhage and cerebellar hemorrhage) patients receiving treatment in four clinical centers (Tangdu Hospital, Ankang Central Hospital, 987 Hospital of PLA Joint Logistic Support Force, and Nuclear Industry 215 Hospital of Shaanxi Province) who meet the screening criteria were invited to participate in this cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 month after onset
  The mortality rate of patients undertook different treatments at 1 month.
Mortality | 6 month after onset
  The mortality rate of patients undertook different treatments at 6 month.
Mortality | 12 month after onset
  The mortality rate of patients undertook different treatments at 12 month.
Neurological Outcome Assessed by modified Rankin Scale (mRS) Score | 1 month after onset
  The neurological function state of patients undertook different treatments at 1 month.
Neurological Outcome Assessed by mRS Score | 6 month after onset
  The neurological function state of patients undertook different treatments at 6 month.
Neurological Outcome Assessed by mRS Score | 12 month after onset
  The neurological function state of patients undertook different treatments at 12 month.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qu, Study Chair — Tang-Du Hospital; Wei Guo, Study Director — Tang-Du Hospital
Locations (1):
- Tandu Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun GC, Chen XL, Hou YZ, Yu XG, Ma XD, Liu G, Liu L, Zhang JS, Tang H, Zhu RY, Zhou DB, Xu BN. Image-guided endoscopic surgery for spontaneous supratentorial intracerebral hematoma. J Neurosurg. 2017 Sep;127(3):537-542. doi: 10.3171/2016.7.JNS16932. Epub 2016 Sep 16. PMID 27636179
- [Background] Broderick J, Connolly S, Feldmann E, Hanley D, Kase C, Krieger D, Mayberg M, Morgenstern L, Ogilvy CS, Vespa P, Zuccarello M; American Heart Association/American Stroke Association Stroke Council; American Heart Association/American Stroke Association High Blood Pressure Research Council; Quality of Care and Outcomes in Research Interdisciplinary Working Group. Guidelines for the management of spontaneous intracerebral hemorrhage in adults: 2007 update: a guideline from the American Heart Association/American Stroke Association Stroke Council, High Blood Pressure Research Council, and the Quality of Care and Outcomes in Research Interdisciplinary Working Group. Circulation. 2007 Oct 16;116(16):e391-413. doi: 10.1161/CIRCULATIONAHA.107.183689. PMID 17938297
- [Background] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637
- [Background] Hanley DF, Thompson RE, Rosenblum M, Yenokyan G, Lane K, McBee N, Mayo SW, Bistran-Hall AJ, Gandhi D, Mould WA, Ullman N, Ali H, Carhuapoma JR, Kase CS, Lees KR, Dawson J, Wilson A, Betz JF, Sugar EA, Hao Y, Avadhani R, Caron JL, Harrigan MR, Carlson AP, Bulters D, LeDoux D, Huang J, Cobb C, Gupta G, Kitagawa R, Chicoine MR, Patel H, Dodd R, Camarata PJ, Wolfe S, Stadnik A, Money PL, Mitchell P, Sarabia R, Harnof S, Barzo P, Unterberg A, Teitelbaum JS, Wang W, Anderson CS, Mendelow AD, Gregson B, Janis S, Vespa P, Ziai W, Zuccarello M, Awad IA; MISTIE III Investigators. Efficacy and safety of minimally invasive surgery with thrombolysis in intracerebral haemorrhage evacuation (MISTIE III): a randomised, controlled, open-label, blinded endpoint phase 3 trial. Lancet. 2019 Mar 9;393(10175):1021-1032. doi: 10.1016/S0140-6736(19)30195-3. Epub 2019 Feb 7. PMID 30739747